CLINICAL TRIAL: NCT03760744
Title: Imaging Biomarkers of Lymphatic Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Manus Donahue, Associate Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 3760744; 1R01NR015079 (NIH)
Record Dates: First submitted 2018-11-28; First posted 2018-11-30 (Actual); Results first posted 2025-10-16 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-09

CONDITIONS: Secondary Lymphedema
Keywords: lymphedema; therapy; swelling; graded negative pressure; complete decongestive therapy
MeSH Terms: conditions — Lymphedema | interventions — carbohydrate-deficient transferrin

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CDT Alone first, then CDT With Negative Pressure (Experimental): Participants randomized into a CDT alone without LymphaTouch for 6 weeks, total of 9 therapy visits (75minutes duration). This is followed by a 6 month washout period, then a second intervention consisting of CDT with LymphaTouch for 6 weeks, total of 9 therapy visits (75minutes duration)
  Interventions: Procedure: CDT with Negative Pressure; Procedure: CDT alone
- CDT With Negative Pressure first, then CDT Alone (Active Comparator): Participants randomized into a CDT with LymphaTouch Negative Pressure for 6 weeks, total of 9 therapy visits (75minutes duration). This is followed by a 6 month washout period, then a second intervention consisting of CDT alone without Negative Pressure for 6 weeks, total of 9 therapy visits (75minutes duration)
  Interventions: Procedure: CDT with Negative Pressure; Procedure: CDT alone

INTERVENTIONS:
Procedure: CDT with Negative Pressure — Complete decongestive therapy (physical therapy conservative intervention of compression, manual lymphatic drainage, skin care and exercises) in conjunction with manual intervention of graded negative pressure application for lymphatic stimulation/ tissue clearance
  Other Names: CDT with LymphaTouch
Procedure: CDT alone — Complete decongestive therapy (physical therapy conservative intervention of compression, manual lymphatic drainage, skin care and exercises) for lymphatic stimulation/ tissue clearance
  Other Names: Complete decongestive therapy without negative pressure

SUMMARY:
Persons with secondary arm and/or upper quadrant lymphedema following cancer therapies commonly are prescribed complete decongestive therapy as a course of management of their lymphedema. The investigators will perform a repeated-measures cross-over trial to test the hypothesis that mobilization of protein enriched hardened tissue using graded negative pressure therapy in conjunction with complete decongestive therapy (CDT) is more effective to standard CDT alone for secondary lymphedema management.

DETAILED DESCRIPTION:
The goal of this work is to apply novel, noninvasive magnetic resonance imaging (MRI) methods for visualizing lymphatic circulation dysfunction to test a fundamental hypothesis about secondary lymphedema conservative decongestive therapy. Breast cancer treatment-related lymphedema (BCRL) arises secondary to surgical axillary lymph node (LN) dissection and irritation, and is a chronic and lifelong condition affecting a high 21.4% of patients receiving common breast cancer therapies. Persons with secondary lymphedema following axillary lymph node removal also include undergoing treatment for other cancers, such as melanoma involving the upper body, necessitating the need for axially lymph node removal.

Improving lymphedema management represents a major clinical need, and emerging efforts focus on improving quality of life through optimizing post-surgical complex decongestive therapy (CDT), and exploring novel pharmacological and surgical procedures. Here, the investigators will perform a repeated-measures cross-over trial to test the hypothesis that mobilization of protein enriched hardened tissue using graded negative pressure therapy in conjunction with complete decongestive therapy (CDT) is more effective to standard CDT alone for secondary lymphedema management. Both of these conservative physical therapy treatments are commonly employed for treatment of secondary lymphedema.

ELIGIBILITY:
Inclusion Criteria:

* Females with a diagnosis of secondary arm and/or upper quadrant lymphedema following cancer treatments

Exclusion Criteria:

* Subjects who have any type of non-MRI compatible bioimplant activated by mechanical, electronic, or magnetic means (e.g., cochlear implants, pacemakers, neurostimulators, biostimulators, electronic infusion pumps, etc.) or are not able to comfortably be able to tolerate the limited fit of the MRI
* Subjects who have any type of ferromagnetic bioimplant that could potentially be displaced.
* Subjects who may have shrapnel embedded in their bodies (such as from war wounds), metal workers and machinists (potential for metallic fragments in or near the eyes).
* Pregnant women will be excluded from the MRI portion of the study only
* Subjects who have open wounds on either ankle or top of foot because of contraindications with placement of electrodes to obtain the L-DEX U400 readings.
* Persons with heart pacemakers.
* Persons with bilateral arm lymphedema (or bilateral risk) or pre-existing lymphedema/edema in the upper body prior to cancer treatments.

Ages: 30 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-01-23 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manus M Donahue, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Donahue PM, Crescenzi R, Scott AO, Braxton V, Desai A, Smith SA, Jordi J, Meszoely IM, Grau AM, Kauffmann RM, Sweeting RS, Spotanski K, Ridner SH, Donahue MJ. Bilateral Changes in Deep Tissue Environment After Manual Lymphatic Drainage in Patients with Breast Cancer Treatment-Related Lymphedema. Lymphat Res Biol. 2017 Mar;15(1):45-56. doi: 10.1089/lrb.2016.0020. PMID 28323572
- [Background] Crescenzi R, Donahue PMC, Hartley KG, Desai AA, Scott AO, Braxton V, Mahany H, Lants SK, Donahue MJ. Lymphedema evaluation using noninvasive 3T MR lymphangiography. J Magn Reson Imaging. 2017 Nov;46(5):1349-1360. doi: 10.1002/jmri.25670. Epub 2017 Feb 28. PMID 28245075

RESULTS

PARTICIPANT FLOW:
Groups:
- CDT Alone First, Then CDT With Negative Pressure: A total of 9 therapy visits (75minutes duration) of CDT alone without LymphaTouch was administered for 6 weeks. After a six month washout participants were brought back in for another 9 therapy visits (75minutes duration) administered over 6 weeks of CDT with Negative Pressure.
  CDT alone: Complete decongestive therapy (physical therapy conservative intervention of compression, manual lymphatic drainage, skin care and exercises) for lymphatic stimulation/ tissue clearance.
  conservative intervention of compression, manual lymphatic drainage, skin care and exercises) for lymphatic stimulation/ tissue clearance CDT with LymphaTouch for 6 weeks, total of 9 therapy visits (75minutes duration) CDT with Negative Pressure: Complete decongestive therapy (physical therapy conservative intervention of compression, manual lymphatic drainage, skin care and exercises) in conjunction with manual intervention of graded negative pressure application for lymphatic stimulation/ tissue clearance.
- CDT With Negative Pressure First, Then CDT Alone: A total of 9 therapy visits (75minutes duration) of CDT alone with LymphaTouch negative pressure was administered for 6 weeks. After a six month washout participants were brought back in for another 9 therapy visits (75minutes duration) administered over 6 weeks of CDT without Negative Pressure.
  CDT alone: Complete decongestive therapy (physical therapy conservative intervention of compression, manual lymphatic drainage, skin care and exercises) for lymphatic stimulation/ tissue clearance.
  conservative intervention of compression, manual lymphatic drainage, skin care and exercises) for lymphatic stimulation/ tissue clearance CDT with LymphaTouch for 6 weeks, total of 9 therapy visits (75minutes duration) CDT with Negative Pressure: Complete decongestive therapy (physical therapy conservative intervention of compression, manual lymphatic drainage, skin care and exercises) in conjunction with manual intervention of graded negative pressure application for lymphatic stimulation/ tissue clearance.
Period: Overall Study
Arm/Group | CDT Alone First, Then CDT With Negative Pressure | CDT With Negative Pressure First, Then CDT Alone
Started | 9 | 9
Completed | 6 | 9
Not Completed | 3 | 0
Not completed — Lost to Follow-up | 3 | 0

BASELINE CHARACTERISTICS:
Population: All participants analyzed were females with unilateral breast-cancer related lymphedema of the upper arm.
Groups:
- CDT Alone First, Then CDT With Negative Pressure: A total of 9 therapy visits (75minutes duration) of CDT alone without LymphaTouch was administered for 6 weeks. After a six month washout period, participants were brought back in for another 9 therapy visits (75minutes duration) administered over 6 weeks of CDT with Negative Pressure.
  CDT alone: Complete decongestive therapy (physical therapy conservative intervention of compression, manual lymphatic drainage, skin care and exercises) for lymphatic stimulation/ tissue clearance.
  CDT with Negative Pressure: Complete decongestive therapy (physical therapy conservative intervention of compression, manual lymphatic drainage, skin care and exercises) in conjunction with manual intervention of graded negative pressure application for lymphatic stimulation/ tissue clearance.
- CDT With Negative Pressure First, Then CDT Alone: A total of 9 therapy visits (75minutes duration) of CDT with LymphaTouch Negative Pressure was administered for 6 weeks. After a six month washout period, participants were brought back in for another 9 therapy visits (75minutes duration) administered over 6 weeks of CDT Alone, without Negative Pressure.
  CDT Alone: Complete decongestive therapy (physical therapy conservative intervention of compression, manual lymphatic drainage, skin care and exercises) for lymphatic stimulation/ tissue clearance.
  CDT with Negative Pressure: Complete decongestive therapy (physical therapy conservative intervention of compression, manual lymphatic drainage, skin care and exercises) in conjunction with manual intervention of graded negative pressure application for lymphatic stimulation/ tissue clearance.
- Total: Total of all reporting groups
Arm/Group | CDT Alone First, Then CDT With Negative Pressure | CDT With Negative Pressure First, Then CDT Alone | Total
Number analyzed (Participants) | 6 | 9 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 8 | 14
  >=65 years | 0 | 1 | 1
Age, Continuous [Median (Full Range); unit: years] | 49.5 [42 to 59] | 51.5 [36 to 75] | 50.5 [36 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 15
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 9 | 15
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 9 | 15

OUTCOME MEASURES:

1. Primary Outcome: Assessing a Change in Bioimpedance Spectroscopy (BIS)
Description: BIS is a noninvasive technology measuring the resistance and reactance of tissue across multiple electrical frequencies using the Impedimed U400 device. By distinguishing ICF from ECF, BIS allows sensitive detection of ECF accumulation, a hallmark of lymphedema. Impedimed's proprietary calculations convert impedance ratios of limbs (involved vs unaffected) into a single output known as LDEX (lymphedema index) with an output normal range of -10 to +10. In situations of overt signs of lymphedema, the LDEX value could be up to 120. This single output value (LDEX) is used in lymphedema research and clinical care to monitor lymphedema progress and response to lymphedema therapy. The LDEX outcome in this study represents the change in LDEX value of the arms from study baseline and at 6-8 weeks following the completion of therapy where a negative value shows a positive response from the therapy intervention by indicating a reduction in the LDEX value.
Time Frame: At baseline and at 6-8 weeks following the completion of therapy
Measure: Mean (Standard Deviation); unit: Change of score on a scale
Units Other Than Participants: affected vs unaffected limbs
Groups:
- CDT Alone: CDT alone without LymphaTouch for 6 weeks, total of 9 therapy visits (75minutes duration)
  CDT alone: Complete decongestive therapy (physical therapy conservative intervention of compression, manual lymphatic drainage, skin care and exercises) for lymphatic stimulation/ tissue clearance
- CDT With Negative Pressure: CDT with LymphaTouch for 6 weeks, total of 9 therapy visits (75minutes duration)
  CDT with Negative Pressure: Complete decongestive therapy (physical therapy conservative intervention of compression, manual lymphatic drainage, skin care and exercises) in conjunction with manual intervention of graded negative pressure application for lymphatic stimulation/ tissue clearance
Arm/Group | CDT Alone | CDT With Negative Pressure
Number analyzed (Participants) | 15 | 15
Number analyzed (affected vs unaffected limbs) | 30 | 30
Change of score on a scale | 1.3 (8) | 1.8 (5.1)

2. Secondary Outcome: Assessing a Change in Quality of Life Via Patient Specific Functional Scale (PSFS)
Description: The Patient Specific Functional Scale (PSFS) was developed as a self-report outcome measure of function that could be used in participants with varying levels of independence. Each participant chose a set of three daily activities and rated the level of ease and comfort with which they could complete them pre and post each intervention.
  Rating scale starts at 0 (unable to perform activity) and goes to goes up to 10 (able to perform activity at the same level as before injury or problem). The closer to 10, the more favorable the number is.
Time Frame: At baseline (pre-intervention) and at 6-8 weeks following the completion of each therapy (post-intervention)
Measure: Mean (Standard Deviation); unit: PSFS score
Arm/Group | CDT Alone | CDT With Negative Pressure
Number analyzed (Participants) | 15 | 15
PSFS score
  At baseline (Pre-Intervention) | 5.1 (2.0) | 5.0 (1.8)
  at 6-8 weeks following the completion of each therapy (Post-Intervention) | 6.6 (2.5) | 7.0 (1.8)

3. Secondary Outcome: Tissue Dielectric Constant (TDC) Measurement Difference Above the Elbow
Description: TDC measures the skin-to-fat water content in tissues. The location was chosen given the propensity of swelling and discomfort in the area for participant population.
  This measurement compares the TDC value in the affected limb versus the unaffected limb, therefore the closer the TDC measurement difference is to zero, the more favorable the value is.
Time Frame: At baseline (pre-intervention) and at 6-8 weeks following the completion of each therapy ([post intervention )
Population: While participants started in different groups, all 15 analyzed participants went through both arms of the study after a washout period. This number represents all participants who completed both arms of the study.
Measure: Mean (Standard Deviation); unit: TDC % change
Units Other Than Participants: affected limb versus the unaffected limb
Arm/Group | CDT Alone | CDT With Negative Pressure
Number analyzed (Participants) | 15 | 15
Number analyzed (affected limb versus the unaffected limb) | 30 | 30
TDC % change
  At Baseline (Pre-Intervention) | 9.8 (10.8) | 9.4 (9.7)
  6-8 weeks following the completion of each therapy (Post-Intervention) | 8.9 (9.5) | 4.8 (5.8)

ADVERSE EVENTS:
Time Frame: 2 years, 4 months.
Arm/Group | CDT Alone | CDT With Negative Pressure
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-07-07): https://cdn.clinicaltrials.gov/large-docs/44/NCT03760744/Prot_SAP_000.pdf